CLINICAL TRIAL: NCT02671266
Title: Effect of Intranasal Oxytocin on Social Cognition
Brief Title: Oxytocin Administration in BDD and OCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2014P001777
Record Dates: First submitted 2016-01-12; First posted 2016-02-02 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Body Dysmorphic Disorder; Obsessive-compulsive Disorder
Keywords: Oxytocin; Body dysmorphic disorder; Obsessive-compulsive disorder
MeSH Terms: conditions — Body Dysmorphic Disorders; Obsessive-Compulsive Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin, Then Placebo (Experimental): Participants will first receive a nasal spray containing the hormone oxytocin (24 IU, 3 puffs per nostril). After a one-week washout period, participants will come back to the clinic and receive a placebo nasal spray (containing all of the same ingredients as the oxytocin spray minus the active oxytocin ingredient).
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo, Then Oxytocin (Experimental): Participants will first receive a placebo nasal spray containing a matching formulation as the oxytocin spray (without the active oxytocin ingredient). After a one-week washout period, participants will come back to the clinic and receive an oxytocin nasal spray (24 IU, 3 puffs per nostril).
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin nasal sprays will be self-administered in the presence of a study nurse. The dose is 24 IU (3 puffs per nostril, 4 IU per puff) of Syntocinon nasal spray.
  Other Names: Syntocinon (Novartis Switzerland)
Drug: Placebo — Placebo nasal sprays will be self-administered in the presence of a study nurse. The sprays will contain all of the same ingredients as the Syntocinon spray minus the active oxytocin ingredient.
  Other Names: Matching placebo formulation

SUMMARY:
The purpose of the current study is to investigate the effect of an acute administration of intranasal oxytocin, relative to placebo, on social cognitive impairments among individuals with body dysmorphic disorder and obsessive-compulsive disorder, compared to healthy controls.

DETAILED DESCRIPTION:
Despite the development of efficacious pharmacologic and psychological treatments body dysmorphic disorder (BDD), treatment outcome data suggest that there is still considerable room for improvement. A closer examination of biological mechanisms underlying psychopathology may help uncover mechanisms to target during intervention and thereby provide a novel approach to treatment. Given that the neuropeptide, oxytocin, is involved in the regulation of a variety of social and cognitive dimensions, including emotion recognition and social attentional processing, there are direct implications regarding its role in the development of such deficits among individuals with BDD. The current study therefore aims to investigate the effect of oxytocin administration on social cognitive impairments in BDD and a related disorder, OCD. Twenty treatment-seeking male and female outpatients with BDD, 20 individuals with OCD, and 20 healthy participants will be assigned to receive an oxytocin and placebo nasal spray one week apart. During each visit, subjects will complete a series of tasks to measure emotion recognition, attentional biases, interpretive biases, and trust behavior. Importantly, these findings may show that a single administration of oxytocin may alter social cognitive processes thought to maintain BDD, and ultimately inform treatments for BDD.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-seeking adult males and females ≥ 18 years of age
* Meets DSM-IV criteria for principal BDD (for BDD group) or principal OCD (for OCD group), as determined by Structured Clinical Interview for DSM-IV (SCID) diagnostic interview
* For females only: must be taking low-dose oral contraceptive pills, as defined by monophasic pills containing <50 mcg ethinyl estradiol
* For healthy volunteers only: does not meet current DSM-IV diagnosis of any Axis I disorder

Exclusion Criteria:

* Participants in the BDD group will be excluded if they have a comorbid diagnosis of OCD and participants in the OCD group will be excluded if they have a comorbid diagnosis of BDD.
* Current diagnosis of schizophrenia, psychotic disorder, bipolar disorder, substance abuse or substance dependence. All other Axis I comorbidities will be permitted to foster the accrual of a clinically relevant sample.
* Significant nasal pathology (e.g., atrophic rhinitis, history of hypophysectomy, recurrent nosebleeds)
* Smokers who smoke ≥ 15 cigarettes daily
* Serious medical illnesses
* Active homicidal or suicidal ideation
* Concurrent use of psychotropic medications
* Steroid or hormone use (except low-dose oral contraceptive pills for females, which is allowed)
* For females only: positive urine pregnancy test and use of high dose estrogen/progestin pills (low dose estrogen/progestin oral contraceptives will be allowed due to stability of hormone levels during active phase)
* For healthy volunteers only: any current DSM-IV Axis I disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fang, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital/Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 20 | 21
BDD Participants | 9 | 9
OCD Participants | 2 | 3
Healthy Participants | 8 | 8
Completed | 19 | 20
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.20 (8.90) | 27.05 (7.00) | 27.12 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 17 | 21 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 14 | 28
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
BDD-YBOCS [Mean (Standard Deviation); unit: units on a scale] — The Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS) is a 12-item clinician administered measure that is designed to assess body dysmorphic disorder symptom severity. Total scores are reported. Total scores range from 0 (least severe) to 48 (most severe). Population: BDD-YBOCS was a clinician-administered measure only administered to patients with body dysmorphic disorder.
  units on a scale
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 25.11 (5.13) | 24.89 (3.55) | 24.89 (4.19)
BABS [Mean (Standard Deviation); unit: units on a scale] — The Brown Assessment of Beliefs Scale (BABS) is a clinician-administered measure designed to assess degree of insight and conviction of beliefs. Total scores are reported. Total scores range from 0 (excellent insight) to 24 (lacks insight, delusional). Population: BABS was a clinician-administered measure that was administered to patients with body dysmorphic disorder and obsessive compulsive disorder.
  units on a scale
    number analyzed (Participants) | 11 | 12 | 23
    (all) | 12.73 (5.82) | 11.17 (3.41) | 11.91 (4.67)

OUTCOME MEASURES:

1. Primary Outcome: Emotion Recognition Questionnaire
Description: This questionnaire includes 48 items for 2 conditions- a self-referent and other-referent condition. Scores are reported for each condition (self-referent or other-referent) reflecting the number of correct responses. Scores range from 0 (least accurate) to 24 (most accurate) for each condition of the questionnaire.
Time Frame: 45 minutes post nasal spray administration
Population: Data reported for BDD and healthy control participants who completed at least one drug visit. There was one patient in the oxytocin first arm who did not complete second placebo drug visit. OCD group was excluded from analyses due to difficulties with recruitment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Number analyzed (Participants) | 17 | 17
score on a scale
  BDD oxytocin- self-referent: number analyzed (Participants) | 9 | 10
  BDD oxytocin- self-referent | 18.67 (3.16) | 17.00 (6.41)
  BDD placebo- self-referent: number analyzed (Participants) | 9 | 10
  BDD placebo- self-referent | 17.00 (3.64) | 16.40 (6.38)
  BDD oxytocin- other-referent: number analyzed (Participants) | 9 | 10
  BDD oxytocin- other-referent | 18.00 (2.40) | 18.30 (6.77)
  BDD placebo- other-referent: number analyzed (Participants) | 9 | 10
  BDD placebo- other-referent | 18.44 (2.96) | 16.40 (6.15)
  HC oxytocin- self-referent: number analyzed (Participants) | 9 | 8
  HC oxytocin- self-referent | 15.67 (6.00) | 17.13 (3.76)
  HC placebo- self-referent: number analyzed (Participants) | 8 | 8
  HC placebo- self-referent | 15.88 (6.64) | 18.88 (3.83)
  HC oxytocin- other-referent: number analyzed (Participants) | 9 | 8
  HC oxytocin- other-referent | 14.78 (5.74) | 16.25 (6.90)
  HC placebo- other-referent: number analyzed (Participants) | 8 | 8
  HC placebo- other-referent | 16.00 (6.52) | 17.88 (3.36)

2. Secondary Outcome: Interpretation Questionnaire
Description: This questionnaire includes 33 ambiguous scenarios, representing 3 conditions: BDD threat scenarios, social anxiety threat scenarios, and general threat scenarios. Each item involves 3 possible thoughts that may come to mind in the scenarios which reflect positive, negative, and neutral interpretations. Participants will be asked to rate the likelihood of having each of the thoughts on a scale of 0 (very unlikely) to 4 (very likely). Total scores are reported for negative threat interpretations for each of the 3 conditions (BDD threat, social anxiety threat, general threat), with scores ranging from 0 (very unlikely) to 44 (very likely).
Time Frame: At least 45 minutes post nasal spray administration
Population: One participant (who received oxytocin first) misunderstood the IQ so was excluded from analysis. One subject who received oxytocin first missed the second placebo drug visit. Another subject who received placebo first accidentally did not receive the Interpretation Questionnaire due to administration error. OCD group was excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Number analyzed (Participants) | 17 | 17
score on a scale
  Oxytocin BDD- BDD threat: number analyzed (Participants) | 8 | 8
  Oxytocin BDD- BDD threat | 24.88 (8.51) | 26.75 (13.50)
  Oxytocin BDD- SA threat: number analyzed (Participants) | 8 | 8
  Oxytocin BDD- SA threat | 27.25 (4.06) | 33.25 (16.29)
  Oxytocin BDD- Gen threat: number analyzed (Participants) | 8 | 8
  Oxytocin BDD- Gen threat | 20.88 (8.48) | 22.38 (6.46)
  Placebo BDD- BDD threat: number analyzed (Participants) | 8 | 9
  Placebo BDD- BDD threat | 21.88 (10.03) | 28.78 (9.01)
  Placebo BDD- SA threat: number analyzed (Participants) | 8 | 9
  Placebo BDD- SA threat | 25.75 (7.76) | 31.11 (6.37)
  Placebo BDD- Gen threat: number analyzed (Participants) | 8 | 9
  Placebo BDD- Gen threat | 19.88 (8.13) | 24.33 (7.86)
  Oxytocin HC- BDD threat: number analyzed (Participants) | 8 | 8
  Oxytocin HC- BDD threat | 10.13 (5.94) | 8.50 (9.09)
  Oxytocin HC- SA threat: number analyzed (Participants) | 8 | 8
  Oxytocin HC- SA threat | 13.38 (5.55) | 12.90 (9.58)
  Oxytocin HC- Gen threat: number analyzed (Participants) | 8 | 8
  Oxytocin HC- Gen threat | 16.75 (6.50) | 15.38 (9.13)
  Placebo HC- BDD threat: number analyzed (Participants) | 7 | 8
  Placebo HC- BDD threat | 7.71 (4.31) | 7.88 (5.59)
  Placebo HC- SA threat: number analyzed (Participants) | 7 | 8
  Placebo HC- SA threat | 15.86 (5.11) | 12.88 (7.85)
  Placebo HC- Gen threat: number analyzed (Participants) | 7 | 8
  Placebo HC- Gen threat | 19.41 (4.82) | 13.63 (8.45)

3. Secondary Outcome: Engagement Towards and Disengagement From Threat Cues in a Spatial Cueing Task
Description: The outcome measures are response latencies (in milliseconds) on engagement and disengagement trials for disgust, happy, and neutral cue types. Longer response latencies reflect more sustained attention.
Time Frame: At least 45 minutes post nasal spray administration
Population: Data reported for BDD and HC participants who completed at least one drug visit. One HC patient in the oxytocin first arm did not complete second placebo visit. Another HC patient in the placebo first arm had missing data from the placebo visit due to administrative error. OCD group was excluded from analyses due to difficulties with recruitment.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Number analyzed (Participants) | 16 | 17
milliseconds
  BDD Oxytocin Happy Engagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Happy Engagement | 636.56 (66.07) | 689.32 (282.68)
  BDD Oxytocin Happy Disengagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Happy Disengagement | 624.08 (78.21) | 581.47 (67.98)
  BDD Oxytocin Neutral Disengagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Neutral Disengagement | 626.80 (74.58) | 594.96 (92.18)
  BDD Oxytocin Neutral Engagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Neutral Engagement | 649.77 (65.46) | 737.74 (361.07)
  BDD Oxytocin Disgust Disengagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Disgust Disengagement | 622.30 (77.45) | 607.09 (111.39)
  BDD Oxytocin Disgust Engagement: number analyzed (Participants) | 9 | 9
  BDD Oxytocin Disgust Engagement | 674.00 (95.03) | 603.94 (83.59)
  BDD Placebo Happy Engagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Happy Engagement | 587.86 (57.84) | 718.41 (401.92)
  BDD Placebo Happy Disengagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Happy Disengagement | 627.45 (106.07) | 610.25 (95.03)
  BDD Placebo Neutral Disengagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Neutral Disengagement | 590.84 (55.10) | 604.59 (62.14)
  BDD Placebo Neutral Engagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Neutral Engagement | 626.99 (116.93) | 614.46 (79.94)
  BDD Placebo Disgust Disengagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Disgust Disengagement | 604.24 (63.82) | 601.19 (66.31)
  BDD Placebo Disgust Engagement: number analyzed (Participants) | 9 | 9
  BDD Placebo Disgust Engagement | 593.57 (52.72) | 625.31 (119.00)
  HC Oxytocin Happy Engagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Happy Engagement | 622.08 (75.20) | 984.01 (452.85)
  HC Oxytocin Happy Disengagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Happy Disengagement | 634.15 (80.27) | 881.50 (270.97)
  HC Oxytocin Neutral Engagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Neutral Engagement | 656.64 (120.41) | 871.63 (336.02)
  HC Oxytocin Neutral Disengagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Neutral Disengagement | 644.85 (137.26) | 781.01 (231.04)
  HC Oxytocin Disgust Disengagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Disgust Disengagement | 613.12 (72.78) | 834.81 (219.30)
  HC Oxytocin Disgust Engagement: number analyzed (Participants) | 7 | 8
  HC Oxytocin Disgust Engagement | 620.73 (75.60) | 826.90 (208.97)
  HC Placebo Happy Engagement: number analyzed (Participants) | 6 | 7
  HC Placebo Happy Engagement | 593.97 (73.17) | 811.25 (200.97)
  HC Placebo Happy Disengagement: number analyzed (Participants) | 6 | 7
  HC Placebo Happy Disengagement | 576.44 (78.04) | 919.46 (268.07)
  HC Placebo Neutral Disengagement: number analyzed (Participants) | 6 | 7
  HC Placebo Neutral Disengagement | 575.38 (108.46) | 774.14 (150.24)
  HC Placebo Neutral Engagement: number analyzed (Participants) | 6 | 7
  HC Placebo Neutral Engagement | 571.02 (84.09) | 847.44 (182.60)
  HC Placebo Disgust Disengagement: number analyzed (Participants) | 6 | 7
  HC Placebo Disgust Disengagement | 603.58 (106.17) | 896.73 (238.16)
  HC Placebo Disgust Engagement: number analyzed (Participants) | 6 | 7
  HC Placebo Disgust Engagement | 560.64 (52.51) | 864.02 (215.64)

4. Secondary Outcome: Amount of Initial Monetary Transfer During Trust Game
Description: Participants will have the decision of sending between 0 to 10 game dollars to another participant, without any expectation of monetary return. This initial investment amount will serve as a measure of trust, with a transfer of 0 game dollars indicating no trust and a transfer of 10 game dollars indicating maximum trust.
Time Frame: At least 45 minutes post nasal spray administration
Population: Sample includes BDD and healthy control participants who completed at least one drug visit. OCD group was excluded from analysis due to difficulties with recruitment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Number analyzed (Participants) | 17 | 17
units on a scale
  Oxytocin BDD- Game 1: number analyzed (Participants) | 9 | 9
  Oxytocin BDD- Game 1 | 6.11 (2.67) | 7.67 (2.50)
  Placebo BDD- Game 1: number analyzed (Participants) | 9 | 9
  Placebo BDD- Game 1 | 7.11 (2.33) | 8.00 (2.50)
  Oxytocin BDD- Game 2: number analyzed (Participants) | 9 | 9
  Oxytocin BDD- Game 2 | 7.22 (2.33) | 6.89 (3.51)
  Placebo BDD- Game 2: number analyzed (Participants) | 9 | 9
  Placebo BDD- Game 2 | 5.22 (3.35) | 8.00 (2.50)
  Oxytocin HC- Game 1: number analyzed (Participants) | 8 | 8
  Oxytocin HC- Game 1 | 6.25 (2.49) | 7.75 (2.19)
  Placebo HC- Game 1: number analyzed (Participants) | 7 | 8
  Placebo HC- Game 1 | 7.71 (2.06) | 5.50 (3.12)
  Oxytocin HC- Game 2: number analyzed (Participants) | 8 | 8
  Oxytocin HC- Game 2 | 7.88 (1.64) | 6.88 (2.75)
  Placebo HC- Game 2: number analyzed (Participants) | 7 | 8
  Placebo HC- Game 2 | 8.29 (1.38) | 5.50 (3.12)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during an approximately two hour period after participant inhaled the nasal spray until completion of the experimental tasks.
Description: Adverse events data were collected by a nurse using a symptom checklist.
Groups:
- Oxytocin: Participants will first receive a nasal spray containing the hormone oxytocin (24 IU, 3 puffs per nostril). After a one-week washout period, participants will come back to the clinic and receive a placebo nasal spray (containing all of the same ingredients as the oxytocin spray minus the active oxytocin ingredient).
  Oxytocin: Oxytocin nasal sprays will be self-administered in the presence of a study nurse. The dose is 24 IU (3 puffs per nostril, 4 IU per puff) of Syntocinon nasal spray.
- Placebo: Participants will first receive a placebo nasal spray containing a matching formulation as the oxytocin spray (without the active oxytocin ingredient). After a one-week washout period, participants will come back to the clinic and receive an oxytocin nasal spray (24 IU, 3 puffs per nostril).
  Placebo: Placebo nasal sprays will be self-administered in the presence of a study nurse. The sprays will contain all of the same ingredients as the Syntocinon spray minus the active oxytocin ingredient.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 15/34 | 17/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=34) | Placebo (N=33)
Feeling drowsy or sleepy (Nervous system disorders) | 12 (12) | 11 (11)
Feeling of calmness or euphoria (Nervous system disorders) | 6 (6) | 6 (6)
Difficulty sitting still (Nervous system disorders) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Trouble concentrating (Nervous system disorders) | 4 (4) | 2 (2)
Blurred vision (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety or depression (Nervous system disorders) | 3 (3) | 2 (2)
Dry mouth/throat (Nervous system disorders) | 2 (2) | 3 (3)
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lightheadedness (Nervous system disorders) | 2 (2) | 4 (4)
Poor memory (Nervous system disorders) | 0 (0) | 2 (2)
Tremors or shakiness (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT02671266/Prot_SAP_000.pdf